CLINICAL TRIAL: NCT04754360
Title: Cut-off Values of 6-min Walk Test and Sit-to-stand Test for Determining Symptom Burden and Functional Impairment in Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Melih Zeren, Assist. Prof. Dr., Izmir Bakircay University
Other Study IDs: bakircaymzeren01
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
Keywords: Symptomatology; Functional impairment; Exercise capacity; 6-min walk test; Sit-to-stand test; Cut-off value
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial fibrillation: Adult patients with atrial fibrillation
  Interventions: Other: Evaluation of functional impairment; Other: Evaluation of pulmonary function; Other: Evaluation of quality of life; Other: Evaluation of physical activity level

INTERVENTIONS:
Other: Evaluation of functional impairment — Symptom burden and functional impairment will be evaluated with EHRA Score, 6-min walk test and 30-second sit-to-stand test
Other: Evaluation of pulmonary function — Pulmonary function will be evaluated using basic spirometry and respiratory pressure meter.
Other: Evaluation of quality of life — Quality of life will be evaluated using Short Form-36 Questionnaire.
Other: Evaluation of physical activity level — Physical activity level will be evaluated using International Physical Activity Questionnaire Short Form

SUMMARY:
Cut-off values indicating higher symptom burden and impairment in health status in 6-min walk test and 30-second sit-to-stand test in patients with atrial fibrillation will be determined in the study.

DETAILED DESCRIPTION:
The 6-min walk test (6MWT) is the most used field test for measuring functional impairment in cardiopulmonary patients. However, to be able to objectively interpret 6MWT of a patient with specific chronic condition, the distance walked in 6MWT should be compared to either a healthy control group or a cut-off value that was specifically determined for that population. Such cut-off values are present for 6MWT in several cardiopulmonary diseases including COPD (350 m), heart failure (200 m) and pulmonary hypertension (400 m) for identifying patients with high mortality, poor prognosis and/or poor health status, but there is no cut-off value determined for atrial fibrillation (AF). The European Heart Rhythm Association (EHRA) score is a practical measure for assessing symptom burden and functional impairment caused by AF-related symptoms. While EHRA class 1 indicates asymptomatic patients, EHRA class 2, 3 and 4 indicates higher severities of symptom burden and functional impairment. Primary aim of this study is to determine a cut-off value in 6MWT for discriminating between the asymptomatic and symptomatic AF patients according to EHRA classification. In addition, a cut-off value for 30-second sit-to-stand test will be determined in these patients as well, since sit-to-stand tests have gained a lot of interest in the recent literature for practically evaluating functional status in various cardiopulmonary conditions.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of paroxysmal, persistant or permanent atrial fibrillation

Exclusion Criteria:

* Diagnosis of heart failure or any chronic respiratory disease
* Recent coronary bypass surgery
* Previous heart valve surgery
* Rheumatic valvular heart disease
* Recent acute myocardial infarction
* Having a pacemaker

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
The European Heart Rhythm Association (EHRA) score | At baseline
  Functional impairment and symptom burden of the patients will be determined according to The European Heart Rhythm Association (EHRA) score. While EHRA class 1 indicates asymptomatic patients, EHRA class 2, 3 and 4 indicates higher severities of symptom burden and functional impairment, respectively.
6-min walk distance | At baseline
  Distance walked in six minutes will be recorded. Test will be conducted according to the guideline of American Thoracic Society (ATS).
Number of repetitions in 30-second sit-to-stand test | At baseline
  Participants will be asked to perform sit-to-stand maneuver as fast as possible for 30 seconds and the number of completed repetitions will be recorded.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | At baseline
  FVC will be measured using basic spirometry according to the guideline of European Respiratory Society (ERS)
Forced Expiratory Volume in 1 second (FEV1) | At baseline
  FEV1 will be measured using basic spirometry according to the guideline of European Respiratory Society (ERS)
Peak Expiratory Flow (PEF) | At baseline
  PEF will be measured using basic spirometry according to the guideline of European Respiratory Society (ERS)
Maximum inspiratory pressure (MIP) | At baseline
  MIP will be measured using electronic mouth pressure meter according to the guideline of European Respiratory Society (ERS)
Maximum expiratory pressure (MEP) | At baseline
  MEP will be measured using electronic mouth pressure meter according to the guideline of European Respiratory Society (ERS)
Short Form-36 | At baseline
  Short Form-36 questionnaire will be used to measure quality of life.
International Physical Activity Questionnaire - Short Form | At baseline
  International Physical Activity Questionnaire - Short Form will be used to measure physical activity level

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Institute of Cardiology, Istanbul, Turkey (Türkiye)